CLINICAL TRIAL: NCT02202889
Title: Improving Bone Health in Adolescence Through Targeted Behavioral Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: University of Hawaii (Other); Arizona State University (Other); University of California, Davis (Other); University of Nevada, Las Vegas (Other); Ohio State University (Other); Southern Illinois University (Other)
Responsible Party: Principal Investigator, Dennis A. Savaiano, Professor and Associate Provost, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00-52102-9696
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Bone Development; Dietary Adequacy
Keywords: Adolescents; Bone mass; Calcium; Perceived milk intolerance; lactose maldigestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Adequate Calcium Today — A school-randomized behavioral intervention study called the Adequate Calcium Today (ACT) project was conducted in sixth grade classrooms located in six states (Arizona, California, Hawaii, Indiana, Nevada, and Ohio).

SUMMARY:
School based educational intervention to educate on bone health among Hispanic, Asian or non-Hispanic white girls between 10-13 years with end points of knowledge gained, calcium intake and bone density in . The hypothesis was that the educational program would increase knowledge, improve dairy food and calcium consumption and enhance bone health in this population. A secondary hypothesis was that lactose maldigestion would be an impediment to improved dairy food consumption.

DETAILED DESCRIPTION:
A targeted behavioral intervention to improve calcium intake and bone mass was conducted at middle schools in 6 states. The primary outcomes of bone mass and dietary calcium were assessed among Asian, Hispanic, or non-Hispanic white girls between 10 -13 y. Lactose maldigestion (LM) was determined by a breath hydrogen test (BHT). Perceived milk intolerance (PMI) and calcium intake were assessed by questionnaires and bone mineral content (BMC) was determined by dual energy X-ray absorptiometry (DXA). Data from 473 girls were used in a multiple linear regression to examine the impact of the intervention while accounting for PMI and LM and adjusting for covariates.

ELIGIBILITY:
Inclusion Criteria:

Middle schools within one-hour driving time of one of the designated DXA measurement sites were eligible to participate in ACT if their student population had a higher proportion of Asian or Hispanic students than the respective state's average. - Girls recruited for evaluation measures were limited to those being at least 75% Asian, Hispanic or non-Hispanic White based on the race/ethnicity of their biological parents.

Exclusion Criteria:

-

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 848 (Actual)
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mineral Content | 18 months
  Baseline, 12 month and 18 month bone mineral content measured
Dietary Calcium | 18 months
  Dietary Calcium intake assessed by food frequency questionnaire

SECONDARY OUTCOMES:
Lactose maldigestion | Baseline
  Measured by breath hydrogen testing

OTHER OUTCOMES:
Perceived lactose intolerance | Baseline
  Measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Savaiano, PhD, Principal Investigator — Purdue University; Carol Boushey, PhD, Principal Investigator — University of Hawaii
Locations (1):
- Purdue University, West Lafayette, Indiana, United States